CLINICAL TRIAL: NCT06969677
Title: Personalized Normative Feedback to Increase HIV Testing Among Adults in Rural Uganda
Brief Title: Personalized Normative Feedback to Increase HIV Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alexander Tsai, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013P000395_4; R01MH125667 (NIH)
Record Dates: First submitted 2025-05-05; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: HIV Testing; HIV Stigma
Keywords: HIV testing; HIV stigma
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Study participants are randomly assigned to be read prompts with personalized normative feedback information with slight changes in content.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- V1: Control Group (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific prompts. The first prompt states the participant's perceived estimate (elicited previously during the survey) of HIV testing rates among single and married people in their village. No other norms-based information is provided.
  Participants are then asked to report their likelihood of getting tested for HIV in the next 12 months, ranging from 1= I will definitely get tested to 5= I will definitely not get tested. Next they are asked to estimate the rate of HIV testing in the next 12 months among men and women in their village, ranging from 1 = All or almost all, at least 90% of group to 5= Very few, or no one, for example, less than 10% of group.
  Interventions: Other: Survey questionnaire
- V2: PNF - Descriptive norms only (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific treatments. The second treatment is a survey-based questionnaire with a prompt stating the participant's perceived estimate (elicited previously during the survey) of HIV testing rates among single and married people in their village. Participants are then provided with the true rates of HIV testing among men and women in their village, along with information that these rate are consistent across demographic groups.
  Participants are then asked to report their likelihood of getting tested for HIV in the next 12 months, ranging from 1= I will definitely get tested to 5= I will definitely not get tested. Next they are asked to estimate the rates of HIV testing in the next 12 months among men and women in their village, ranging from 1 = All or almost all, at least 90% of group to 5= Very few, or no one, for example, less than 10% of group.
  Interventions: Other: Survey questionnaire
- V3: PNF - Injunctive norms only (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific treatments. The third treatment is a survey-based questionnaire with a prompt stating the participant's perceived estimate (elicited previously during the survey) of HIV testing rates among single and married people in their village. Participants are then provided with information about the true rates of HIV stigma in their village.
  Participants are then asked to report their likelihood of getting tested for HIV in the next 12 months, ranging from 1= I will definitely get tested to 5= I will definitely not get tested. Next they are asked to estimate the rate of HIV testing in the next 12 months among men and women in their community, ranging from 1 = All or almost all, at least 90% of group to 5= Very few, or no one, for example, less than 10% of group.
  Interventions: Other: Survey questionnaire
- V4: PNF - Descriptive and injunctive norms (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific treatments. The fourth treatment is a survey-based questionnaire with a prompt stating the participant's perceived estimate (elicited previously during the survey) of HIV testing rates among single and married people in their village. Participants are then provided with information about the true rates of both HIV testing and HIV stigma in their village.
  Participants are then asked to report their likelihood of getting tested for HIV in the next 12 months, ranging from 1= I will definitely get tested to 5= I will definitely not get tested. Next they are asked to estimate the rate of HIV testing in the next 12 months among men and women in their community, ranging from 1 = All or almost all, at least 90% of group to 5= Very few, or no one, for example, less than 10% of group.
  Interventions: Other: Survey questionnaire

INTERVENTIONS:
Other: Survey questionnaire — Each version of the questionnaire has similar questions about personal HIV testing intentions and perceived norms about other men and women's HIV testing intentions. The content of the prompt presented prior to the questions varies based on treatment arm.
  This version does not provide any normative feedback information.
  Arms: V1: Control Group
Other: Survey questionnaire — Each version of the questionnaire has similar questions about personal HIV testing intentions and perceived norms about other men and women's HIV testing intentions. The content of the prompt presented prior to the questions varies based on treatment arm.
  This version provides personalized normative feedback with descriptive norms information about local HIV testing rates.
  Arms: V2: PNF - Descriptive norms only
Other: Survey questionnaire — Each version of the questionnaire has similar questions about personal HIV testing intentions and perceived norms about other men and women's HIV testing intentions. The content of the prompt presented prior to the questions varies based on treatment arm.
  This version provides personalized normative feedback with injunctive norms information about local HIV stigma rates.
  Arms: V3: PNF - Injunctive norms only
Other: Survey questionnaire — Each version of the questionnaire has similar questions about personal HIV testing intentions and perceived norms about other men and women's HIV testing intentions. The content of the prompt presented prior to the questions varies based on treatment arm.
  This version provides personalized normative feedback with descriptive and injunctive norms information about both local HIV testing rates and local HIV stigma rates.
  Arms: V4: PNF - Descriptive and injunctive norms

SUMMARY:
Randomized trial to measure the effect of personalized normative feedback about local HIV testing rates and local rates of HIV-related stigma on self-reported HIV testing intentions and perceptions about others' HIV testing intentions.

DETAILED DESCRIPTION:
HIV testing is a vital step in identifying and treating HIV. Research in rural Uganda reveals underestimation of community HIV testing rates and overestimation of HIV-related stigma among adults. At the same time, perceived norms (i.e., estimated rates regardless of their accuracy) are associated with personal HIV testing behavior and personal HIV-related attitudes.

This study employs a randomized controlled trial to evaluate how providing accurate information about local descriptive (i.e., behavioral) norms and local injunctive (i.e., attitudinal) norms affect HIV testing intentions. Participants are randomly assigned to one of four treatment arms: (1) they are reminded of what they thought community testing rates were in their village and then receive accurate information about high community testing rates, (2) they are reminded of what they thought local stigma rates were in their village and then receive accurate information about positive community perceptions of persons with HIV, (3) they are reminded of what they thought community testing rates and local stigma rates were in their village and then receive both types of accurate normative information, or (4) they are reminded of what they thought community testing rates were in their village and receive no further information (control group).

The study assesses how providing this type of personalized normative feedback within cohort-based data collection affects personal reports about getting tested for HIV in the next 12 months and how it affects perceptions about how many men and women in the same village will get tested for HIV in the next 12 months. It is hypothesized that providing accurate information about local community testing rates and/or attitudes toward persons with HIV will increase reported personal willingness to get tested (primary outcome) and improve the accuracy of estimated community testing rates in the future (secondary outcome).

ELIGIBILITY:
Inclusion Criteria:

* All adults who consider Nyakabare their primary place of residence and who are capable of providing consent

Exclusion Criteria:

* Minors younger than 18 years of age, with the exception of emancipated minors
* Persons who do not consider Nyakabare Parish their primary place of residence, e.g. persons who happen to be visiting Nyakabare at the time of the survey or who own a home in Nyakabare but spend most of their time outside of the parish
* Persons with psychosis, neurological damage, acute intoxication, or other cognitive impairment (all of which are determined informally in the field by non-clinical research staff in consultation with a supervisor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1300 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Self-reported HIV testing intention in the next 12 months | Baseline (assessed at the time the survey is administered)
  Regarding yourself, how likely are you to go get tested for HIV in the next 12 months? (single item)

SECONDARY OUTCOMES:
Self-reported perception of HIV testing among men in one's village | Baseline (assessed at the time the survey is administered)
  How many of these men do you think will go get tested for HIV in the next 12 months? (single item)
Self-reported perception of HIV testing among women in one's village | Baseline (assessed at the time the survey is administered)
  How many of these women do you think will go get tested for HIV in the next 12 months? Read all response options audibly, except for refuses/do not know.
  (single item)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Tsai, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No